CLINICAL TRIAL: NCT01156935
Title: Effects of Laugh-yoga Intervention on Mood and Quality of Life Among Oncologic Patients
Brief Title: Effects of Laugh-yoga Intervention on Mood and Quality of Life Among Oncologic Patients in a Oncologic Clinic Setting.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dr. Yossef Brener, Wolfson MC
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 0073-10-WOMC
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Neoplasms
Keywords: Neoplasm; Laugh-Yoga; Mood; Quality of life
MeSH Terms: conditions — Neoplasms

ARMS (1):
- Laugh yoga (Experimental): experimental laugh yoga
  Interventions: Other: Laugh Yoga

INTERVENTIONS:
Other: Laugh Yoga — 1 hour including laugh, respiratory exercises and guided imagination by a group instructor specialized in laugh yoga

SUMMARY:
Previous studies report low levels of mood and of quality of life among cancer patients. Laugh has been proved to improve mood and immune system function. The investigators propose to assess in a prospective randomised case-control study the affects of laugh-yoga intervention on mood levels and quality of life among cancer patients in a cancer clinic. The main hypothesis is that patients in laugh-yoga group will report higher mood and quality o life levels after intervention in comparison with no-intervention group. The second hypothesis is that immune system is the mediator of the effects of laugh-yoga intervention on mood and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* oncologic patients treated in oncologic clinic in Wolfson MC,
* must be able to participate in Laugh Yoga session

Exclusion Criteria:

* psychiatric or cognitive impairment,
* deterioration in physical status,
* treatment discontinuation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaire - QLQ-C30 & Positive-Negative Affect | Participants will fill QLQ-C30 & Positive -Negative Affect will be assessed before intervention and after three laugh - yoga sessions (that is after three weeks)

SECONDARY OUTCOMES:
Blood analysis for WBC, CRP, T&B Lymphocytes | Before intervention and after three laugh-yoga interventions, that is after three weeks.